CLINICAL TRIAL: NCT04470882
Title: Use of Safety Behaviors in Exposure Therapy for Arachnophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Cynthia Lancaster, Assistant Professor, Clinical Psychology, University of Nevada, Reno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1330971-1
Record Dates: First submitted 2019-04-11; First posted 2020-07-14 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Specific Phobia; Arachnophobia; Spider Phobia
Keywords: Exposure therapy; Safety behaviors; Arachnophobia; Spider phobia; Specific phobia
MeSH Terms: conditions — Phobia, Specific; Arachnophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure with faded safety behaviors (Experimental): Exposure therapy will involve three, 10-minute trials in which participants encounter a spider. Participants in this group will wear protective gear during the first two trials, and will remove the protective gear during the last trial.
  Interventions: Behavioral: Exposure with faded safety behaviors
- Exposure without safety behaviors (Active Comparator): Exposure therapy will involve three, 10-minute trials in which participants encounter a spider. Participants in this group will not wear protective gear during any of the exposure therapy trials.
  Interventions: Behavioral: Exposure without safety behaviors
- Exposure with unfaded safety behaviors (Experimental): Exposure therapy will involve three, 10-minute trials in which participants encounter a spider. Participants in this group will wear protective gear during all three exposure therapy trials.
  Interventions: Behavioral: Exposure with unfaded safety behaviors

INTERVENTIONS:
Behavioral: Exposure with faded safety behaviors — Exposure therapy will involve three, 10-minute trials in which participants encounter a spider. Participants in this group will wear protective gear during the first two trials, and will remove the protective gear during the last trial.
  Arms: Exposure with faded safety behaviors
Behavioral: Exposure without safety behaviors — Exposure therapy will involve three, 10-minute trials in which participants encounter a spider. Participants in this group will not wear protective gear during any of the exposure therapy trials.
  Arms: Exposure without safety behaviors
Behavioral: Exposure with unfaded safety behaviors — Exposure therapy will involve three, 10-minute trials in which participants encounter a spider. Participants in this group will wear protective gear during all three exposure therapy trials.
  Arms: Exposure with unfaded safety behaviors

SUMMARY:
This study examines the impact of safety behaviors (i.e., unnecessary protective actions) on outcomes of exposure therapy for spider phobia. Researchers will compare exposure therapy with (a) no safety behaviors, (b) safety behaviors faded toward the end of treatment, and (c) unfaded safety behaviors.

DETAILED DESCRIPTION:
Some studies suggest that safety behaviors might undermine the efficacy of exposure therapy (Powers et al., 2010), whereas other studies suggest that there is no difference in exposure therapy outcomes whether or not safety behaviors are used (Deacon et al., 2010). Mixed findings could be explained by the parameters of safety behaviors use, such as whether they are used throughout the full course of therapy or faded toward the end of therapy. This will be the first study to directly compare the impact of faded and unfaded safety behaviors on exposure therapy outcomes. Specifically, researchers will randomize participants with a fear of spiders to receive exposure therapy (a) without safety behavior use, (b) with faded safety behavior use, and (c) with un-faded safety behavior use. Researchers will compare each condition's impact on fear reduction and on the tolerability/acceptability of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Displays sufficiently high fear of spiders, as indicated by responses on (a) a self report questionnaire (the Fear of Spiders Questionnaire) at prescreening, and (b) Behavioral Avoidance Tests at baseline

Exclusion Criteria:

* younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Behavioral approach test (treatment context) - behavioral outcome | Change from baseline up to 4 weeks later (through follow up assessment)
  Participants will approach a live, non-poisonous tarantula, placed on the floor, at the opposite end of the room. The participant will walk toward the spider during this test. The test is over when the participant has reached the hardest step that they can complete at that time.
  During this BAT, investigators will assess fear response behaviorally by recording the most challenging step completed (range, steps 0 -12).
Behavioral approach test (treatment context) - subjective outcome | Change from baseline up to 4 weeks later (through follow up assessment)
  Participants will approach a live, non-poisonous tarantula, placed on the floor, at the opposite end of the room. The participant will walk toward the spider during this test. The test is over when the participant has reached the hardest step that they can complete at that time.
  During this BAT, investigators will assess fear response subjectively by having participants self report their peak fear level (on a 0 to 100 scale).
Behavioral approach test (treatment context) - physiological outcome | Change from baseline up to 4 weeks later (through follow up assessment)
  Participants will approach a live, non-poisonous tarantula, placed on the floor, at the opposite end of the room. The participant will walk toward the spider during this test. The test is over when the participant has reached the hardest step that they can complete at that time.
  During this BAT, investigators will assess fear response physiologically by assessing heart rate variability.
Behavioral approach test (generalization context) - behavioral outcome | Change from baseline up to 4 weeks later (through follow up assessment)
  Participants will approach a live, non-poisonous tarantula, placed in a clear tank on a table, at the opposite end of the room. The test is over when the participant has reached the hardest step that they can complete at that time. Steps include walking toward the spider and lowering one hand into the tank.
  During this BAT, investigators will assess fear response behaviorally by recording the most challenging step completed (range, steps 0-21).
Behavioral approach test (generalization context) - subjective outcome | Change from baseline up to 4 weeks later (through follow up assessment)
  Participants will approach a live, non-poisonous tarantula, placed in a clear tank on a table, at the opposite end of the room. The test is over when the participant has reached the hardest step that they can complete at that time. Steps include walking toward the spider and lowering one hand into the tank.
  During this BAT, investigators will assess fear response subjectively by having participants self report their peak fear level (on a 0 to 100 scale).
Behavioral approach test (generalization context) - physiological outcome | Change from baseline up to 4 weeks later (through follow up assessment)
  Participants will approach a live, non-poisonous tarantula, placed in a clear tank on a table, at the opposite end of the room. The test is over when the participant has reached the hardest step that they can complete at that time. Steps include walking toward the spider and lowering one hand into the tank.
  During this BAT, investigators will assess fear response physiologically by assessing heart rate variability.
Fear of Spiders Questionnaire (FSQ) | Change from baseline up to 4 weeks later (through follow up assessment)
  Self-report rating scale in which participants rate the extent that they agree with a number of statements that are representative of having a fear of spiders. Sum total scores will be calculated (range 0-108). Higher scores indicate more severe symptom levels.
Spider Phobia Beliefs Questionnaire (SBQ) | Change from baseline up to 4 weeks later (through follow up assessment)
  Self-report rating scale assessing the level to which the participant believes a number of cognitions/thoughts commonly associated with spider phobia. An overall average rating will be calculated (range 0-100). Higher average scores indicate greater belief in spider phobic cognitions.
Armfield and Mattiske Disgust Questionnaire (AMDQ) | Change from baseline up to 4 weeks later (through follow up assessment)
  Self-report questionnaire assessing feelings of disgust associated with spiders. Sum total scores will be calculated (range 0-48). Higher scores indicate more severe spider-related disgust.
Anxiety Disorders Interview Schedule for DSM-5 (ADIS-5) | Change from baseline up to 4 weeks later (through follow up assessment)
  Participants will be given a structured interview to identify whether they meet diagnostic criteria for specific phobia. Responses will be coded dichotomously (yes = has diagnosis; no = no diagnosis).

SECONDARY OUTCOMES:
Treatment Acceptability/Adherence Scale (Modified version) | Measured just prior to beginning a one-session treatment
  Self-report questionnaire assessing the participant's perceptions regarding treatment acceptability and willingness to adhere to treatment procedures. Sum total scores will be calculated (range 10-70). Higher scores indicate greater acceptability/adherence.
Treatment Acceptability/Adherence Scale (Modified version) | Measured immediately after completing a one-session treatment
  Self-report questionnaire assessing the participant's perceptions regarding treatment acceptability and willingness to adhere to treatment procedures. Sum total scores will be calculated (range 10-70). Higher scores indicate greater acceptability/adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

REFERENCES:
- [Background] Powers MB, Smits JA, Telch MJ. Disentangling the effects of safety-behavior utilization and safety-behavior availability during exposure-based treatment: a placebo-controlled trial. J Consult Clin Psychol. 2004 Jun;72(3):448-54. doi: 10.1037/0022-006X.72.3.448. PMID 15279528
- [Background] Deacon BJ, Sy JT, Lickel JJ, Nelson EA. Does the judicious use of safety behaviors improve the efficacy and acceptability of exposure therapy for claustrophobic fear? J Behav Ther Exp Psychiatry. 2010 Mar;41(1):71-80. doi: 10.1016/j.jbtep.2009.10.004. Epub 2009 Oct 24. PMID 19892318